CLINICAL TRIAL: NCT01842425
Title: Changes in Body- and Liver-composition During Low Calorie Diet in Morbidly Obese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, DEdholm, MD, Uppsala University
Other Study IDs: MR-LCD2
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
Keywords: Liver volume; Gastric bypass; Magnetic resonance imaging
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two serum samples from each patient at each examination. Biopsies of subcutananeous fat and visceral fat, approximately 1 mililiter each, taken during laparoscopic gastric bypass surgery
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine what changes occur in body- and liver-composition during four weeks of low calorie diet in morbidly obese females

DETAILED DESCRIPTION:
Preoperative weight loss prior to laparoscopic gastric bypass is desirable as this reduces liver volume and thus facilitates the visualization of the gastro-esophageal junction. Weight loss is often achieved through low-calorie diet (LCD); however the ideal duration of LCD treatment is unknown.

Morbidly obese female patients awaiting laparoscopic gastric bypass are recruited. They are, as all our patients, treated during four weeks with LCD to achieve a decrease in liver size. During this period they are examined on day 0, 3, 7, 14 and 28 after commencing LCD.

At each evaluation, body composition is assessed through bioelectric impedance analysis (BIA), liver volume and intrahepatic fat through magnetic resonance imaging. A questionnaire regarding quality of life and LCD-related symptoms is administered as well. At surgery two samples of subcutaneous fat and one sample of omental fat is taken.

We do not assign patients to different treatments, instead all are treated similarly according to our routine preoperative regimen.

ELIGIBILITY:
Inclusion Criteria:

* Awaiting laparoscopic gastric bypass
* Residing near Uppsala

Exclusion Criteria:

* Weight above 140 kg
* Metal implants such as pacemaker or intracerebral clips
* Failure to understand or comply with study protocol

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Morbidly obese females awaiting laparoscopic gastric bypass surgery
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Liver volume | From baseline to after four weeks

SECONDARY OUTCOMES:
Composition of body fat in subcutaneous and omental fat | At surgery
Changes in body composition | Baseline to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Edholm, MD, Principal Investigator — Department of Surgery
Locations (1):
- Department of surgery, Akademiska sjukhuset, Uppsala, Sweden